CLINICAL TRIAL: NCT06526559
Title: The Evaluation of Barbed Sutures Versus Non-barbed Sutures in Minimally Invasive Dismembered Pyeloplasty. A Prospective Randomized Controlled Study.
Brief Title: Barbed Versus PGA Sutures in Minimally Invasive Dismembered Pyeloplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Fakhry Makki, Urology Specialist in Cairo University Hospital, Principal investigator, MD Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD-439-2023
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Pelvi-Ureteric Obstruction
Keywords: Pyeloplasty; Dismembered pyeloplasty; Laparoscopic pyeloplasty; Robot-assisted pyeloplasty; Barbed suture
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization is done using a web-based platform, group assignment will only be known to the surgeon (care provider). It would be concealed to the patient, investigator, and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Barbed suture group (Experimental): Pyeloplasty done using barbed absorbable sutures
  Interventions: Device: Barbed suture
- PGA group (Active Comparator): Pyeloplasty done using conventional PGA (Polyglactin) sutures
  Interventions: Device: PGA suture

INTERVENTIONS:
Device: Barbed suture — Use of two absorbable barbed sutures for each arm in the ureteropelvic anastomosis in minimally invasive dismembered pyeloplasty
  Other Names: V-Loc
  Arms: Barbed suture group
Device: PGA suture — Use of two absorbable polyglactin sutures for each arm in the ureteropelvic anastomosis in minimally invasive dismembered pyeloplasty
  Other Names: Vicryl
  Arms: PGA group

SUMMARY:
The main goals of this trial is to study the feasibility and safety of using barbed sutures compared to the conventional PGA (Polyglactin) sutures in minimally invasive dismembered pyeloplasty. The main questions in using barbed sutures would be:

1. Is it safe with similar post-operative outcomes?
2. Does it have any significant complications?
3. Is it easier to handle intra-operatively?

DETAILED DESCRIPTION:
Minimally invasive surgeries for pelviureteric junction obstruction have become more popular in the past decade than open surgery. This is to decrease the morbidity for patients and attain better patient satisfaction especially for having a significantly smaller incisions compared to open flank and midline abdominal incisions.

Minimally invasive surgery is a term used to describe surgeries that would spare the patient a long incision and hence spares him also the pain and risk of wound infection associated with it. In this study the investigators will focus only on laparoscopy and robot-assisted surgeries.

Pelviureteric junction obstruction is a disease that is not uncommon with an incidence of 1 in 1000-1500. Although usually it is diagnosed in the pediatric population, it is not uncommon in adults. PUJO (Pelviureteric junction obstruction) could have it's impact on the patient's quality of life as if it is not treated it could decrease the split glomerular filtration rate due to impaired drainage. It also could present with secondary renal stones, pain, recurrent upper urinary tract infection, fever and urosepsis.

Management of PUJO (Pelviureteric junction obstruction) starts with the proper assessment of the patient regarding his age and careful history taking and physical examination, evaluation of laboratory investigations such as urine culture and sensitivity, serum creatinine, total leucocytic count. Also, evaluation of the pelviabdominal ultrasound, intravenous pyelography, and diuretic renogram.

Treatment of PUJO (Pelviureteric junction obstruction) ranges from active surveillance, endopyelotomy and ureteral stenting, and pyeloplasty whether it is open, laparoscopic or robot-assisted.

Traditionally, absorbable polyglactin sutures is used for dismembered pyeloplasty. Yet recently barbed sutures have gained popularity within urologists especially in minimally invasive surgeries.

Barbed knotless uni-directional sutures have the benefit of being knotless and evenly distributes tension so there is no need for the assistant to follow the surgeon and stretch the suture, this significantly decreases the operative time and frees the assistant's port to be able to do other steps.

Barbed sutures have been well established in other surgical fields such as bariatric surgery, gynecology, and skin closure previously, and recently it has been populated in the urological community especially in the vesicourethral anastomosis in Radical prostatectomy.

Sparse yet promising articles have been published regarding the use of barbed sutures in pyeloplasty which could change the way surgeons approach the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 undergoing robotic or laparoscopic dismembered pyeloplasty
* History of dietls' crisis (Fever, pain) in a pelviureteric junction obstructed kidney
* Decrease in glomerular filtration rate in a pelviureteric junction obstructed kidney

Exclusion Criteria:

* Contraindications for laparoscopy or robotic surgery as pulmonary obstructive or restrictive disease, and poor cardiovascular fitness
* Uncontrolled diabetes mellitus
* Morbid obesity
* History of multiple major abdominal surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Time difference for suture completion | 12 months (Intra-operative data)
  Mean difference of time taken in minutes between each group
Difference in complications rate | 18 months (Post-operative data)
  Mean difference in complications rate between both groups
Drain output post-operative | 12 months (Early post-operative data)
  Mean difference in total drain output between both groups

SECONDARY OUTCOMES:
Difference in total operative time | 12 months (Intra-operative data)
  Mean difference in total operative time post-operative
Difference in hospitalization time | 12 months (Early post-operative data)
  Mean difference in hospitalization time
Failure rate | 18 months (Late post-operative data)
  Difference in number of patients who needed redo pyeloplasty or any auxiliary procedures

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghoneima, MD, Study Chair — Professor - Urology Department - Reconstructive Urology Unit Cairo University; Ayman Kassem, MD, Study Director — Assistant Professor - Urology Department - Oncology Unit - Cairo University; Mohammed Elghorably, Study Director — Lecturer - Urology Department - King Fahd Hospital - Cairo University; Ahmed Sharawy, MD, Study Director — Lecturer - Urology Department - King Fahd Hospital - Cairo University
Locations (1):
- Cairo University Kasr AlAiny Hospitals Urology Department 17B, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publishing minimum after 18 months for whenever needed

REFERENCES:
- [Result] Shah HN, Nayyar R, Rajamahanty S, Hemal AK. Prospective evaluation of unidirectional barbed suture for various indications in surgeon-controlled robotic reconstructive urologic surgery: Wake Forest University experience. Int Urol Nephrol. 2012 Jun;44(3):775-85. doi: 10.1007/s11255-011-0075-y. Epub 2011 Nov 6. PMID 22057590
- [Result] Anand S, Jukic M, Krishnan N, Pogorelic Z. Barbed Versus Non-Barbed Suture for Pyeloplasty via the Minimally Invasive Approach: A Systematic Review and Meta-Analysis. J Laparoendosc Adv Surg Tech A. 2022 Oct;32(10):1056-1063. doi: 10.1089/lap.2021.0868. Epub 2022 May 12. PMID 35549514
- [Result] Giri V, Yadav SS, Tomar V, Jha AK, Garg A. Retrospective comparison of outcomes of laparoscopic pyeloplasty using barbed suture versus nonbarbed suture: A single-center experience. Urol Ann. 2019 Oct-Dec;11(4):410-413. doi: 10.4103/UA.UA_123_15. PMID 31649463